CLINICAL TRIAL: NCT04760249
Title: The Impact of a Dedicated Sedation Team on the Incidence of Complications in Paediatric Procedural Analgosedation
Brief Title: A Dedicated Sedation Team for Paediatric Procedural Sedation
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: CAST-01
Record Dates: First submitted 2021-02-07; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Sedation Complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
At a tertiary care university hospital a specialized interdisciplinary team of paediatric anaesthesiologists and paediatric intensivists was established for providing analgosedation for diagnostic and therapeutic procedures. The aim of the present study was to analyse the incidence and risk factors of adverse events during procedural sedation performed by the Children's Analgosedation Team (CAST).

DETAILED DESCRIPTION:
At a tertiary care university hospital a dedicated Children's Analgosedation Team (CAST) performs all procedural sedations in children outside the operating room. Often patient age, comorbidities and procedures involving the airway are considered risk factors for adverse events, but previous studies investigating adverse events did not involve implementation of a specialised sedation team. Medical records of all children receiving procedural sedation by the CAST were reviewed for the incidence of adverse events. A bivariate analysis as well as an analysis of variance using type II Wald chi-square tests were conducted for identifying potential risk factors for adverse Events.

ELIGIBILITY:
Inclusion Criteria:

* Children (age 0-20 years) receiving procedural sedation
* Procedural sedation performed by the Children's Analgosedation Team

Exclusion Criteria:

* Missing medical records
* Procedural sedation not performed by the Children's Analgosedation Team

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children from 1 day to 20 years
Sampling Method: Non-Probability Sample
Enrollment: 784 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | From the beginning of sedation (administration of 1. sedation drug) until the end of sedation (patient regained consciousness), assessed up to 6 hours
  Respiratory, hemodynamic, and other adverse events

SECONDARY OUTCOMES:
Incidence of serious adverse events | From the beginning of sedation (administration of 1. sedation drug) until the end of sedation (patient regained consciousness), assessed up to 6 hours
  Aspiration, vomiting/regurgitation, desaturation < 90% for > 30sec, hypotension < 50% of baseline, laryngospasm, thorax rigidity, unplanned admission to Paediatric Intensive Care Unit (PICU), cardiac arrest, and death
Age | At the beginning of sedation (administration of 1. sedation drug)
  Patient age in month
Sex | At the beginning of sedation (administration of 1. sedation drug)
  Male or female
American Society of Anesthesiology (ASA) status | At the beginning of sedation (administration of 1. sedation drug)
  ASA physical status I / II / III / IV
Date of sedation | At the beginning of sedation (administration of 1. sedation drug)
  Date as YEAR/MONTH/DAY
Category of the primary diagnosis | At the beginning of sedation (administration of 1. sedation drug)
  Diagnosis that prompted the need for the procedure, categorized according to the subspecialty (hematology/oncology, nephrology, hepatology, gastroenterology, metabolic medicine, neurology, pulmonology, cardiology)
Type and dose of sedative | From the beginning of sedation (administration of 1. sedation drug) until the end of sedation (patient regained consciousness), assessed up to 6 hours
  Propofol or Midazolam in mg kg-1
Type and dose of analgesic | From the beginning of sedation (administration of 1. sedation drug) until the end of sedation (patient regained consciousness), assessed up to 6 hours
  Esketamine in mg kg-1 or remifentanil in µg kg-1 min-1
Upper respiratory tract infection (URI) | At the beginning of sedation (administration of 1. sedation drug)
  Signs of runny nose and/or cough